CLINICAL TRIAL: NCT04786899
Title: Sleep & Postoperative Delirium in Hispanic/ Latino Patients After Cardiothoracic Surgery
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Elizabeth Mahanna Gabrielli, Assistant Professor of Anesthesiology, University of Miami
Other Study IDs: 20200942
Record Dates: First submitted 2021-03-03; First posted 2021-03-08 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Delirium in Old Age; Sleep Disturbance; Circadian Rhythm Sleep Disorder
MeSH Terms: conditions — Parasomnias; Sleep Disorders, Circadian Rhythm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hispanic/Latino patients undergoing cardiothoracic surgery: Observational study of patients scheduled for cardiothoracic surgery as part of standard of care. Patients will be followed up to 30 days prior to surgery and up to 7 days after surgery or hospital discharge, whichever is sooner. Patients preoperative sleep patterns and postoperative delirium will be followed.

SUMMARY:
The purpose of this research is to study pre-operative sleep problems and delirium in Hispanic/Latino patients after heart and lung surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Self identify as Hispanic/Latino or preferred language as Spanish
2. Undergoing scheduled elective and urgent cardiothoracic surgery
3. 50 years of age and older

Exclusion Criteria:

1. Inability to consent
2. preferred language other than English, Spanish or Portuguese
3. emergency surgery
4. anticipated discharge < 48 hours
5. Individuals < 50 years of age
6. Pregnant women
7. Prisoners

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hispanic/Latino patients scheduled for cardiothoracic surgery at the University of Miami.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2021-02-12 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative delirium in Hispanic/Latino patients after cardiothoracic surgery | Up to 7 days post surgery.
  Delirium will be assessed using the Confusion Assessment Method.

SECONDARY OUTCOMES:
Percentage of participants with preoperative sleep disturbance | Up to 7 days before surgery
  Sleep disturbance as measured by actigraphy data using a wrist-actigraph
Pittsburgh Sleep Quality Index (PSQI) score | baseline
  Pittsburgh Sleep Quality Index (PSQI) score with overall score ranging from 0-21, where lower scores indicate a higher sleep quality.
Insomnia Severity Index (ISI) score | baseline
  Insomnia Severity Index (ISI) score has a total score ranging from 0 to 28, with higher scores signifying greater insomnia severity.
Epsworth Sleepiness scale (ESS) score | baseline
  Epsworth Sleepiness scale (ESS) score has a total score ranging from 0 to 24, with a higher score indicating greater daytime sleepiness.
STOP-BANG Score | baseline
  STOP-BANG Score has a total score ranging from 0 to 8, with higher scores indicating a higher risk of obstructive sleep apnea.
Percentage of patients with risk allele of the melatonin receptor single nucleotide polymorphism. | baseline
  Assess from blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Mahanna Gabrielli, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No